CLINICAL TRIAL: NCT06593847
Title: Multisite Virtual Reality Intervention for Speech Anxiety
Acronym: ETC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of Texas at Austin (Other); Curtin University (Other); Erasmus University Rotterdam (Other); National University of Singapore (Other); Southern Illinois University (Other); Tufts University (Other); The University of New South Wales (Other); University of Western Sydney (Other); University of Arizona (Other); The University of Hong Kong (Other); Philipps Universität Marburg (Unknown); Albright College (Unknown); Utrecht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7565E
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Public Speaking; Speech Anxiety
MeSH Terms: conditions — Speech; Glossophobia

STUDY DESIGN:
Intervention Model Description: Single session VR-based exposure therapy
Masking Description: Participants are blind to the study hypothesis and outcomes are assessed by participant self-report.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive or Negative Mood Induction via film clips (Other): VR exposure is the only intervention, but the VR intervention is conducted following either positive or negative mood induction.
  Interventions: Behavioral: Single-session VR exposure intervention

INTERVENTIONS:
Behavioral: Single-session VR exposure intervention — VR exposure is the only intervention, but the VR intervention is conducted following either positive or negative mood induction.

SUMMARY:
Exposure-based cognitive behavior therapy is an efficacious treatment for speech anxiety and has been delivered effectively in a virtual reality (VR) environment. The present multicenter study (conducted through the Exposure Therapy Consortium) is designed to evaluate whether trait versus state positive affectivity is a more effective predictor of exposure therapy outcomes. Further, the investigators will examine whether the predictive significance of trait positive affectivity can be accounted for by examination of baseline levels of self-efficacy, hope, and optimism.

DETAILED DESCRIPTION:
The goal of this multicenter clinical trial is to examine predictors of VR exposure therapy outcomes for college students with public speaking anxiety following a positive or negative mood induction. The overarching aim of the present study is to evaluate whether trait versus state positive affectivity is a more effective predictor of exposure therapy outcomes. Further, the investigators will examine whether the predictive significance of trait positive affectivity can be accounted for by examination of baseline levels of self-efficacy, hope, and optimism. State affect is manipulated at an experimental level with affect induction procedures; trait positive affectivity is measured at baseline.

The study involves three phases: (1) initial screening, (2) in-person assessment and brief exposure intervention for a subset of participants with elevated public speaking anxiety, and (3) a one-week follow-up assessment conducted online. Students who choose to participate and screen high on a public speaking anxiety scale will be assigned to a positive or negative mood induction condition prior to undergoing VR-based exposure therapy. Public speaking and social anxiety outcomes are measured immediately post-intervention and one week later. The one-week follow-up assessment represents the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of 18 - 70 years of age
* Current student at a participating University
* Ability to read English to provide informed consent
* Familiarity with a computer keyboard and mouse or a touch screen device (e.g. phone, tablet).
* For Phase 2: speech anxiety scale score of ≥ 18 on the Personal Report of Communication Apprehension, Public Speaking Subscale (PRCA-PS)

Exclusion Criteria:

* Previous participation (i.e., no participant may take the survey more than once).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1542 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Public Speaking Anxiety | One week follow-up assessment
  Assessed using the Personal Report of Communication Apprehension, Public Speaking Subscale (PRCA-PS). Scores range from 6 to 30, with higher scores associated with higher public speaking anxiety.

SECONDARY OUTCOMES:
Valence | One week follow-up assessment
  Self-report measure of how participant feels about having to give a speech
Assessed using the Social Phobia Inventory (SPIN) | One week follow-up assessment
  Assessed using the Social Phobia Inventory (SPIN). Scores range from 0-68, with higher scores indicating greater social phobia.
Public Speaking Anxiety | Post-treatment assessment immediately after the intervention
  Assessed using the Personal Report of Communication Apprehension, Public Speaking Subscale (PRCA-PS). Scores range from 6 to 30, with higher scores associated with higher public speaking anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Otto, PhD, Principal Investigator — Boston University
Locations (13):
- United States (6):
  - University of Arizona, Tucson, Arizona
  - Southern Illinois University, Carbondale, Illinois
  - Tufts University, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Albright College, Reading, Pennsylvania
  - University of Texas at Austin, Austin, Texas
- Australia (3):
  - Western Sydney University, Penrith, New South Wales
  - University of New South Wales, Sydney, New South Wales
  - Curtin University, Bently, Western Australia
- University of Hong Kong, Pokfulam, Hong Kong, China
- Philipps-Universität Marburg, Marburg, Hesse, Germany
- Netherlands (2):
  - Erasmus University, Rotterdam, South Holland
  - Utrecht University, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Data will be posted on the Open Science Foundation site.
Supporting Information: Study Protocol
Time Frame: Within one year of study completion.
Access Criteria: Via request to the Exposure Therapy Consortium
URL: https://exposure.la.utexas.edu/

REFERENCES:
- See also: Exposure Therapy Consortium — https://exposure.la.utexas.edu/